CLINICAL TRIAL: NCT04144777
Title: Efficacy of Solarplast for Health and Oxidative Stress, A Randomized, Double-Blind, Placebo-Controlled Study
Brief Title: Efficacy of Solarplast for Health and Oxidative Stress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Deerland Enzymes (Industry)
Collaborators: Kennesaw State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: SP19
Record Dates: First submitted 2019-10-23; First posted 2019-10-30 (Actual); Last update posted 2021-02-15 (Actual); Status verified 2019-10

CONDITIONS: Oxidative Stress; Healthy Aging; Skin Health
Keywords: Smokers; Prediabetes; Cognitive Health
MeSH Terms: conditions — Prediabetic State

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): Subjects will be administered one daily dose of Solarplast (100mg), in a capsule, for 45 days.
  Interventions: Dietary Supplement: Solarplast
- Placebo (No Intervention): Subjects will be administered one daily dose of maltodextrin (100mg), in a capsule, for 45 days.

INTERVENTIONS:
Dietary Supplement: Solarplast — Subjects will take one capsule of Solarplast (100mg) daily for 45 days.
  Arms: Treatment

SUMMARY:
Solarplast is a unique mixture of antioxidant enzymes and single antioxidant molecules that are capable of attack oxidants that cause damage to the cells in the human body and cause premature aging. This mechanism may provide protection from stress, such as free radicals, heat, infection, as well as reduce inflammation and participate in the repair mechanism of the intestinal tract. Participants will consume Solarplast, or placebo, for 45 days with blood draws at day-0 and -45 in order to assess antioxidant capacity.

DETAILED DESCRIPTION:
Solarplast is currently sold on the market, which is a unique mixture of antioxidant enzymes and single antioxidant molecules that attack oxidants through chaperone activity. Chaperones, are naturally occurring proteins that assist the non-covalent folding/unfolding and the assembly/disassembly of other macromolecular structures and can provide stability and restore function of many unfolded proteins. Chaperones may provide protection from stress, such as free radicals, heat, infection, as well as reduce inflammation and participate in the repair mechanism of the intestinal tract. Solarplast is derived from Spinach (Spinacia oleracea), a leafy green vegetable of high nutritional value grown and consumed worldwide. Spinach is rich in iron, vitamin A, riboflavin, and lutein, a carotenoid that acts as a natural antioxidant protecting the body from toxins and free radicals. The potential mechanistic role of Solarplast consists of serving an antioxidant role against peroxyl radicals, hydroxyl radicals, peroxynitrite, super oxide anion, singlet oxygen, among others. Additionally, Solarplast contains photosynthetic complexes with high concentrations of ATP, NADPH, ADP, AMP, NADP, niacin, B12, adenine, and ribose. Therefore, this naturally occurring antioxidant supplement may provide the components required to scavenge free radicals and mitigate oxidative stress with no harmful side effects.

The purpose of this study is to determine the antioxidant and health effects of Solarplast in 40 healthy human subjects, 20 smokers, and 20 pre-diabetics; both male and female (n=80). An equal number of males and females will be recruited for the project. Only participants between the ages of 18 and 55 will be recruited for this research. Smokers and pre-diabetics are known to have increased oxidative stress; therefore, these two populations are being included in this research.

A single capsule of Solarplast containing 100 mg (1 x 10^6 light converting units (LCU)) is to be consumed once a day per participant for a total of 45 days, following pre-screening and enrollment (detailed below). Twenty healthy (of the 40 healthy) human subjects will be used as control subjects and consume a placebo (maltodextrin - 100 mg).

A medical doctor will approve the enrollment (Dr. Karleena Tuggle) of all participants and oversee this clinical trial.

Participants will be asked to visit the laboratory (KSU Human Performance Laboratory) on 2 separate occasions for blood draws by a CITI approved/IRB approved research team member trained in phlebotomy under the supervision of Dr. VanDusseldorp.

ELIGIBILITY:
Inclusion Criteria:

* Healthy smokers
* Healthy non-smokers
* Prediabetics (elevated fasting blood glucose of 100-125mg/dL).

Exclusion Criteria:

* No specific pulmonary disease
* No medication or specifically any inhaled bronchodilators or corticosteroids.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2019-07-15 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
Oxidative Stress | 45 days
  Analyze change in reactive oxygen species obtained from blood from baseline to 45 days using reactive oxygen species testing kits
Blood glucose | 45 days
  Analyze change in fasting blood glucose obtained from blood from baseline to 45 days using metabolic panel
Change in skin health using questionnaires | 45 days
  Analyze skin health using questionnaires
Change in joint pain using questionnaires | 45 days
  Analyze change in joint pain using questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Trisha VanDusseldorp, PhD, Principal Investigator — Kennesaw State University
Locations (1):
- Kennesaw State University, Kennesaw, Georgia, United States

IPD SHARING:
Plan to Share IPD: No